CLINICAL TRIAL: NCT00907816
Title: Concurrent Electronic Order Entry Variation Reporting Impact on Ordering
Brief Title: Concurrent Electronic Order Entry Variation Reporting Impact on Ordering Behavior
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Jeffrey B. Weilburg MD; Associate Medical Director, Mass General Physicians Organization, Massachusetts General Hospital, Boston, MA
Other Study IDs: PHRC Study 2009P-000611
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Behavior
Keywords: this study does not look at patient conditions
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intervention: PCPs at MGH who receive display of utilization and quality during computer order entry
- control

SUMMARY:
Display of information regarding utilization and quality to primary care physicians as they use our computer based system to order radiologic imaging (CT, MR, etc) will reduce unnecessary imaging.

ELIGIBILITY:
Inclusion Criteria:

* PCPs at MGH with patient panel > 99 loyal patients

Exclusion Criteria:

* PCPs at MGH with patient panel < 99 loyal patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PCPs at MGH
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Health status adjusted utilization of imaging by each PCP in the intervention group, compared to themselves before intervention, and as a group to the control group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B. Weilburg, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States